CLINICAL TRIAL: NCT02723071
Title: An Open-label, Multicentre, Dose-escalating Phase I/II Trial of 3-weekly Ocrelizumab in Patients With Follicular Non-Hodgkin's Lymphoma (NHL)
Brief Title: A Study of Ocrelizumab in Participants With Follicular Non-Hodgkin's Lymphoma (NHL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO18414; 2004-004110-17 (EudraCT Number)
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ocrelizumab

ARMS (3):
- Cohort A: Ocrelizumab 200 mg/m^2 (Experimental): Participants will receive a total of 8 infusions of ocrelizumab 200 milligram per square meter (mg/m^2) given at intervals of 3 weeks, until disease progression or unacceptable toxicity.
  Interventions: Drug: Ocrelizumab
- Cohort B: Ocrelizumab 375 mg/m^2 (Experimental): Participants will receive a total of 8 infusions of ocrelizumab 375 mg/m^2 given at intervals of 3 weeks, until disease progression or unacceptable toxicity.
  Interventions: Drug: Ocrelizumab
- Cohort C: Ocrelizumab 375/750 mg/m^2 (Experimental): Participants will receive first infusion of ocrelizumab 375 mg/m^2 followed by 7 infusions of 750 mg/m^2 given at intervals of 3 weeks, until disease progression or unacceptable toxicity.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Participants will receive a total of 8 intravenous (IV) infusions of ocrelizumab given at intervals of 3 weeks, until disease progression or unacceptable toxicity.
  Other Names: RO4964913

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics, and anti-tumor efficacy of ocrelizumab in participants with progressive follicular NHL.

ELIGIBILITY:
Inclusion Criteria:

* Follicular NHL
* Documented history of response, or stable disease more than 6 months in duration, to a rituximab-containing regimen that was the last treatment before enrollment in the study
* No evidence of hepatitis B or C

Exclusion Criteria:

* Prior monoclonal antibody therapy other than rituximab, anti-cancer vaccine, or radioimmunotherapy for cancer
* History of severe allergic or anaphylactic reaction to humanized or murine monoclonal antibodies, or known sensitivity or allergy to murine products
* Major nondiagnostic surgery within 4 weeks of Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose-limiting Toxicity (DLT) | first cycle (3-week cycle) of Cohort A, Cohort B, and Cohort C

SECONDARY OUTCOMES:
Progression-free Survival According to the International Workshop to Standardize Response Criteria for NHL | Day 1, after 4 and 8 cycles of therapy (12 and 24 weeks after study entry) until disease progression/relapse, or death, whichever occurred first (overall up to approximately 2.75 years)
Event-free Survival According to the International Workshop to Standardize Response Criteria for NHL | Day 1, after 4 and 8 cycles of therapy (12 and 24 weeks after study entry) until disease progression/relapse, or death, whichever occurred first (overall up to approximately 2.75 years)
Area Under the Plasma Concentration-Time Curve From Time 0 to Day 28 (AUC0-28) of Ocrelizumab | Pre-infusion (0-2 hours); 30 minutes post infusion on Day 1 of Cycles 1 to 8 (Cycle length = 21 days); Days 2, 8, and 15 of Cycle 1 (Cohorts A, B), Cycle 2 (Cohort C), and Cycle 8 (Cohorts A, B, C); Days 176, 190, 204, 259, 322, 357, 539
Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity AUC(0-inf) of Ocrelizumab | Pre-infusion (0-2 hours); 30 minutes post infusion on Day 1 of Cycles 1 to 8 (Cycle length = 21 days); Days 2, 8, and 15 of Cycle 1 (Cohorts A, B), Cycle 2 (Cohort C), and Cycle 8 (Cohorts A, B, C); Days 176, 190, 204, 259, 322, 357, 539
Percentage of Participants With Overall Response According to the International Workshop to Standardize Response Criteria for NHL | Day 1, after 4 and 8 cycles of therapy (12 and 24 weeks after study entry) until disease progression/relapse, or death, whichever occurred first (overall up to approximately 2.75 years)
Maximum Plasma Concentration (Cmax) of Ocrelizumab | Pre-infusion (0-2 hours); 30 minutes post infusion on Day 1 of Cycles 1 to 8 (Cycle length = 21 days); Days 2, 8, and 15 of Cycle 1 (Cohorts A, B), Cycle 2 (Cohort C), and Cycle 8 (Cohorts A, B, C); Days 176, 190, 204, 259, 322, 357, 539
Systemic Clearance (CL) of Ocrelizumab | Pre-infusion (0-2 hours); 30 minutes post infusion on Day 1 of Cycles 1 to 8 (Cycle length = 21 days); Days 2, 8, and 15 of Cycle 1 (Cohorts A, B), Cycle 2 (Cohort C), and Cycle 8 (Cohorts A, B, C); Days 176, 190, 204, 259, 322, 357, 539
Steady State Volume of Distribution (Vss) of Ocrelizumab | Pre-infusion (0-2 hours); 30 minutes post infusion on Day 1 of Cycles 1 to 8 (Cycle length = 21 days); Days 2, 8, and 15 of Cycle 1 (Cohorts A, B), Cycle 2 (Cohort C), and Cycle 8 (Cohorts A, B, C); Days 176, 190, 204, 259, 322, 357, 539
Terminal Elimination Half-Life (t1/2) of Ocrelizumab | Pre-infusion (0-2 hours); 30 minutes post infusion on Day 1 of Cycles 1 to 8 (Cycle length = 21 days); Days 2, 8, and 15 of Cycle 1 (Cohorts A, B), Cycle 2 (Cohort C), and Cycle 8 (Cohorts A, B, C); Days 176, 190, 204, 259, 322, 357, 539
Number of Participants With Peripheral Blood B-cell Depletion | Week 24, 28 days following the final infusion (Day 176), 9, 18, 24, and 30 months after study entry or until B cell recovery, whichever occurred first (up to approximately 2.75 years)
Number of Participants With Peripheral Blood B-cell Recovery | Week 24, 28 days following the final infusion (Day 176), 9, 18, 24, and 30 months after study entry or until B cell recovery, whichever occurred first (up to approximately 2.75 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- Australia (3):
  - Melbourne
  - Perth
  - Woolloongabba
- Canada (5):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Ottawa, Ontario
  - Toronto, Ontario
- France (5):
  - Créteil
  - Lille
  - Nantes
  - Pierre-Bénite
  - Rennes
- Italy (3):
  - Bergamo
  - Roma
  - Torino
- Sweden (4):
  - Huddinge
  - Lund
  - Malmo
  - Umeå
- Switzerland (3):
  - Bern
  - Geneva
  - Lugano